CLINICAL TRIAL: NCT02813447
Title: Safety of Anti-Depressant for Chronic Obstructive Pulmonary Disease
Brief Title: Safety of Anti-Depressant for Chronic Obstructive Pulmonary Disease (SAD-COPD)
Acronym: SAD-COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 hold
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00071349
Record Dates: First submitted 2016-06-13; First posted 2016-06-27 (Estimated); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2021-09

CONDITIONS: COPD; Anxiety; Depression; Stress; Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Depression; Lung Diseases, Interstitial | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pulmonary Rehab + Study Drug (Active Comparator): Subjects randomized into this arm will be given active study drug (sertraline). Subjects will take 25mg tablets by mouth daily starting at visit 1 along with participating in the intensive pulmonary rehab program. Subjects will be assessed at one week intervals +/- 7 days for tolerability and side effects, and if tolerating study drug, the dose will be increased weekly by 25mg over the course of the first four weeks with maximum effective dose of 100mg daily by the end of week four. Subjects will continue this dose over the course of the remaining 8 weeks of the study, while participating in the graduate program of pulmonary rehab.
  Interventions: Drug: Sertraline
- Pulmonary Rehab + Placebo (Placebo Comparator): Subjects randomized to the placebo arm will have the same procedures as described above in the study drug arm with the exception that they will be receiving matched placebo drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline
  Arms: Pulmonary Rehab + Study Drug
Drug: Placebo
  Arms: Pulmonary Rehab + Placebo

SUMMARY:
Objective: Determine whether treatment of perceived stress, anxiety, and depression with anti-depressant therapy improves dyspnea scores, 6-minute walk (6MW) distance and quality of life (QoL) in patients with Chronic Obstructive Pulmonary Disease (COPD) and ILD (Interstitial Lung Disease) undergoing pulmonary rehab.

The study is a prospective, randomized, double-blinded, placebo-controlled study to assess the effect of an SSRI on 6MW, dyspnea scores, and QoL in COPD and ILD patients undergoing pulmonary rehab. Thirty subjects that carry an ICD-9 code diagnosis of COPD and/or ILD and CES-D (Center for Epidemiologic Studies Depression) score of > 16 will be recruited from Duke Pulmonary Rehab.

Multivariable regression models will be constructed to evaluate the relationship between perceived stress, anxiety, and depression with adjustments by race, gender, age, BMI and GOLD score. A multivariable regression model will be constructed to assess whether treatment of perceived stress, depression, and anxiety with antidepressant therapy (sertraline) is an effect modifier on 6MW distance and dyspnea scores in patients with COPD or ILD who are enrolled in pulmonary rehab.

Descriptive statistics will be used to examine the socio-demographic characteristic data. Student t-tests will be performed to assess group differences in continuous data. Categorical variables will be examined using the Pearson's Chi-Squared test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with an ICD-9 code diagnosis of COPD and/or ILD
* Mild, moderate, or severe major depression symptoms based on Center of Epidemiologic Studies Depression (CES-D) score > 16.
* Able to complete informed consent†
* Read and write in English

Exclusion Criteria:

* Current treatment with antidepressants
* Current treatment with anti-psychotics
* Severe physical disability that would interfere with lung assessment
* History of major psychiatric illness, including bipolar disorder, psychoses, and/or severe personality disorder.
* Active suicidal ideations
* Serious cognitive problems (dementia syndrome) or cognitive impairment defined as MMSE < 22
* Recent loss of spouse within 6 weeks of study enrollment.
* History of alcohol or drug dependence in the last 6 months.
* Pregnant women or nursing mothers
* Poorly controlled concomitant conditions that pose additional procedure risk as determined by the investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mathews, MD, Principal Investigator — Duke University
Locations (1):
- Duke Pulmonary Rehabilitation, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulmonary Rehab + Study Drug: Subjects randomized into this arm will be given active study drug (sertraline). Subjects will take 25mg tablets by mouth daily starting at visit 1 along with participating in the intensive pulmonary rehab program. Subjects will be assessed at one week intervals +/- 7 days for tolerability and side effects, and if tolerating study drug, the dose will be increased weekly by 25mg over the course of the first four weeks with maximum effective dose of 100mg daily by the end of week four. Subjects will continue this dose over the course of the remaining 8 weeks of the study, while participating in the graduate program of pulmonary rehab.
  Sertraline
- Pulmonary Rehab + Placebo: Subjects randomized to the placebo arm will have the same procedures as described above in the study drug arm with the exception that they will be receiving matched placebo drug.
  Placebo
Period: Overall Study
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
Started | 6 | 7
Completed | 1 | 5
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in 6MW Distance
Description: Patients will undergo 6-minute walk at visit 1(baseline), visit 4 (after one month of study drug + intensive pulmonary rehab), and visit 6 (week 12).
Time Frame: visit 1(baseline), visit 4 (after one month of study drug + intensive pulmonary rehab), and visit 6 (week 12).
Population: only participants who completed all 3 visits (visits 1, 4, and 6) were included in the analysis.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
Number analyzed (Participants) | 1 | 5
feet
  change from baseline to Visit 4 | -264.00 (0) | 273.20 (103.89)
  change from baseline to Visit 6 | -94.00 (0) | 163.60 (312.50)

2. Primary Outcome: Change in Dyspnea Scores, as Measured by UCSD Medical Center Pulmonary Rehabilitation Program Shortness of Breath Questionnaire (UCSD-SOB)
Description: To monitor changes in dyspnea scores, patients will complete the UCSD Medical Center Pulmonary Rehabilitation Program Shortness of Breath Questionnaire (UCSD-SOB). Participants will complete this at all visits (1-6). The UCSD is a 24-item questionnaire that asks participants to rate themselves from 0 ("Not at all") to 5 ("Maximally or unable to do because of breathlessness"). Scores range from 0-120, with higher scores indicating greater dyspnea.
Time Frame: visit 1(baseline), visit 4 (week 4), visit 6 (week 12)
Population: Participants with data at the indicated time points are included in the analysis. All collected data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
Number analyzed (Participants) | 3 | 4
score on a scale
  Baseline | 62.67 (8.08) | 36.00 (14.33)
  Change from Baseline to Visit 4: number analyzed (Participants) | 2 | 2
  Change from Baseline to Visit 4 | -0.50 (6.36) | 7.50 (26.16)
  Change from Baseline to Visit 6: number analyzed (Participants) | 1 | 1
  Change from Baseline to Visit 6 | 0.00 (0.00) | -14.00 (0.00)

3. Secondary Outcome: Change in Quality of Life, as Measured by Ferrans & Powers Quality of Life Index - Pulmonary Version (QOL)
Description: To monitor changes in quality of life, patients will complete the Ferrans & Powers Quality of Life Index - Pulmonary version (QOL). Scores range from 0 to 30, with higher scores indicating a higher quality of life.
Time Frame: visit 1(baseline), visit 4 (after one month of study drug + intensive pulmonary rehab), and visit 6 (week 12).
Population: Participants with data at the indicated time points are included in the analysis. All collected data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
Number analyzed (Participants) | 6 | 7
score on a scale
  Baseline | 19.23 (5.26) | 20.12 (2.77)
  Change from Baseline to Visit 4: number analyzed (Participants) | 1 | 1
  Change from Baseline to Visit 4 | 4.53 (0.00) | -0.40 (0.00)
  Change from Baseline to Visit 6: number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Perceived Stress, as Measured by General Health Questionnaire-12 (GHQ-12)
Description: To monitor changes in perceived stress, patients will complete the General Health Questionnaire-12 (GHQ-12). Scores range from 0 to 36, with higher scores indicating greater distress.
Time Frame: visit 1(baseline), visit 4 (after one month of study drug + intensive pulmonary rehab), and visit 6 (week 12).
Population: Participants with data at the indicated time points are included in the analysis. All collected data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
Number analyzed (Participants) | 3 | 4
score on a scale
  Baseline | 16.33 (6.51) | 11.50 (5.07)
  GHQ Change from Baseline to Visit 4: number analyzed (Participants) | 2 | 3
  GHQ Change from Baseline to Visit 4 | -2.50 (2.12) | -3.67 (3.79)
  GHQ Change from Baseline to Visit 6: number analyzed (Participants) | 0 | 1
  GHQ Change from Baseline to Visit 6 |  | -7.00 (0.00)

5. Secondary Outcome: Change in Anxiety, as Measured by Hamilton Anxiety and Depression Scale (HADS)
Description: Scores on the HADS range from 0-21, with higher scores indicating more severe of symptoms.
Time Frame: visit 1(baseline), visit 4 (after one month of study drug + intensive pulmonary rehab), and visit 6 (week 12).
Population: Participants with data at the indicated time points are included in the analysis. All collected data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
Number analyzed (Participants) | 3 | 4
score on a scale
  Baseline | 16.67 (6.11) | 11.00 (6.98)
  Change from Baseline to Visit 4: number analyzed (Participants) | 2 | 3
  Change from Baseline to Visit 4 | -6.50 (3.54) | -0.67 (2.08)
  Change from Baseline to Visit 6: number analyzed (Participants) | 1 | 1
  Change from Baseline to Visit 6 | -3.00 (0.00) | -7.00 (0.00)

6. Secondary Outcome: Change in Anxiety, as Measured by the Anxiety Inventory for Respiratory Disease (AIR) Questionnaire
Description: Scores on the Anxiety Inventory for Respiratory Disease (AIR) range from 0-30, with higher scores indicating more symptoms.
Time Frame: visit 1(baseline), visit 4 (after one month of study drug + intensive pulmonary rehab), and visit 6 (week 12).
Population: Participants with data at the indicated time points are included in the analysis. All collected data are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
Number analyzed (Participants) | 0 | 1
score on a scale
  Baseline |  | 15.00 (0.00)
  Visit 4: number analyzed (Participants) | 0 | 0
  Visit 6: number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Pulmonary Rehab + Study Drug | Pulmonary Rehab + Placebo
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pulmonary Rehab + Study Drug (N=6) | Pulmonary Rehab + Placebo (N=7)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pulmonary Rehab + Study Drug (N=6) | Pulmonary Rehab + Placebo (N=7)
nausea, vomiting and jitteriness (Gastrointestinal disorders) | 1 | 0
drowsiness, lethargy and jitteriness (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The data captured was deemed unreliable due to the turnover among study personnel and insufficient personnel to administer the questionnaires accurately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT02813447/Prot_SAP_000.pdf